CLINICAL TRIAL: NCT06684457
Title: Patient Perceived Degree of Empathy Exhibited by Physician Guided, Prompt Engineered, Generative AI Chatbot Designed for Atrial Fibrillation Education
Brief Title: Patient Perceived Empathy of an AI Chatbot for Atrial Fibrillation Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Samir Saba, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY24010018
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation (AF)
Keywords: education; lifestyle modification; atrial fibrillation; generative AI; chatbot; artificial intelligence
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Study design:
  A single center, cross sectional, uncontrolled, open-label, non-randomized, single arm, experimental pilot study using an LLM based prompt-engineered education chatbot, to impart a Q and A format atrial fibrillation education to patients, prior to their first appointment with a cardiologist or a cardiac electrophysiologist. The prompt-engineered chatbot is built on LLM capabilities yet tailored with the help of physician provided, vetted, open source atrial fibrillation educational material as well as empathy enhancing scripts, and simplified language to a 6th-8th grade reading level. The chatbot would be utilized to enhance the patient-provider interaction by providing empathetic education to patients regarding atrial fibrillation, and empower them with the knowledge they would need to ask informed questions during their patient visit. The chatbot will also be able to direct patients to Heart Rhythm Society's open source educational videos for atrial fibrillation (UpBeat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pilot interventional arm (Experimental): Single arm, wherein all consenting participants undergoing interaction with chatbot for atrial fibrillation education.
  Interventions: Behavioral: Atrial Fibrillation Education

INTERVENTIONS:
Behavioral: Atrial Fibrillation Education — Atrial fibrillation education rendered through a generative AI chatbot, using an iPAD. The intervention itself is an approximately 1 hour long interaction with the chatbot or approximately 10 questions about atrial fibrillation, for 1 single interaction.

SUMMARY:
Atrial Fibrillation is a chronic disease with significant health consequences like increased risk of stroke, heart failure, heart attack and death. Educating patients about the disease is important for them to be able to understand the condition better, feel empowered and take an active part in their care plan. AI technology can potentially be used to impart such education. However, doing so with care and empathy is equally important.

Therefore, it is necessary to ensure when AI technology is used to impart education about atrial fibrillation to patients, the humane aspects of the interaction are rigorously tested. This study examines a way to impart atrial fibrillation education through interaction with an AI chatbot, that uses text and links to educational videos. To participate in this study, people need to be age 18 or older and have a history of newly diagnosed atrial fibrillation. Approximately 40 individuals will be asked to take part in this study.

The first step to the study will be reading through, understanding, and signing an informed consent. People who then agree to join the study will have a one-time interaction with the AI chatbot and structured educational material by using an iPad provided to them for the approximately 1 hour duration of the study. People in the study will obtain atrial fibrillation education by typing one by one on the iPad, up to 10 questions about the disease. Answers will include text and links to videos. Before and after atrial fibrillation education, people who join this study will be asked to fill out a survey. The study team will teach patients how to use the iPad and type in questions.

DETAILED DESCRIPTION:
Background:

Atrial fibrillation is a the most common arrhythmic disorder in the United States, with significant morbidity and healthcare cost burden. The number of patients with atrial fibrillation is expected to reach 12.1 million in 2030. AFib related annual incremental healthcare costs were estimated to be $6 to $26 billion based on 2010AF prevalence projections.

Lifestyle modification is one of the four primary pillars of atrial fibrillation care, and patient education is paramount to foster behavioral change. There is also evidence that early rhythm control using medications and ablation therapy can mitigate the overall burden of atrial fibrillation and improve patient quality of life among patients with other cardiovascular risk factors and/or heart failure. However, social determinants of health including health literacy significantly impact patient management, referral practices for procedural interventions, and ultimately patients' clinical outcomes. Anticoagulation prescription for prevention of thromboembolic complications, and adherence to anticoagulation are also known to be correlated with patients' medical literacy and disease awareness. These data point to three important unmet needs. First, there is a need for more robust and intentional patient education to foster behavioral change including lifestyle modification. Second, patient awareness and understanding of the disease is paramount to facilitate anticoagulation adherence and seeking specialist referral which in turn could mitigate AFib related morbidity and healthcare costs. Third, patient education must be delivered in empathetic language, at a (6th-8th) grade reading level, and translated to languages other than English per patient preference.

In that context, LLMs (large language models) such as ChatGPT (Open AI, San Francisco), with built in capabilities for language simplification and translation could play a foundational role in modern medicine. Current data show that LLMs(Chat GPT) are capable of answering patient queries in an empathetic and knowledgeable manner. Data showing improved readability of surgical consent forms simplified using ChatGPT, while maintaining medical information and medicolegal integrity demonstrate the potential of using LLMs for consent processes and shared decision making. However, it is important to note that providing appropriate guardrails to minimize probabilistic guess responses and fine tune the content for accuracy and empathy requires human interaction with the software. The availability of such prompt-engineered technology for patient education could have a profound impact on patient behavior, clinical outcomes and provider-patient relationship.

ELIGIBILITY:
Inclusion criteria:

* Age greater than18 yrs
* Known diagnosis of atrial fibrillation

Exclusion criteria:

* Inability to text/use an electronic device
* Inability to read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Empathy | From enrollment to end of interaction with chatbot, approximately an hour
  Assess patient perceived degree of empathy exhibited by chatbot responses. The degree of empathy will be measured using a pre- and post- chatbot interaction 7 point Likert scale survey, with a higher score suggesting a higher level of perceived empathy. The title of the survey will be "Likert scale based survey for perceived empathy and trust," with the lowest score being 4 and the highest score being 28. Survey form available upon reasonable request.

SECONDARY OUTCOMES:
Knowledge | From enrollment to end of interaction with chatbot, approximately an hour
  Assess knowledge about AFib imparted by chatbot based on patient survey questions. Knowledge will be measured by administering a pre- and post- bot interaction survey, titled "Jessa Atrial Fibrillation Knowledge Questionnaire," with a minimum score of 0 and a maximum score of 16. A higher score reflects that the patient is more knowledgeable about atrial fibrillation. Survey form available upon reasonable request.
Trust | From enrollment to end of interaction with chatbot, approximately an hour
  Assess impact of chatbot interaction on patient perceived trust in the provider. The degree of trust will be measured using a pre- and post- chatbot interaction 7 point Likert scale survey, with a higher score suggesting a higher level of perceived empathy. The title of the survey will be "Likert scale based survey for perceived empathy and trust," with the lowest score being 4 and the highest score being 28. Survey form available upon reasonable request.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Saba, MD, Principal Investigator — UPMC Heart and Vascular Institute
Locations (1):
- UPMC Heart and Vascular Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified IPD may be shared at the discretion of investigators, upon reasonable request.